CLINICAL TRIAL: NCT02665390
Title: Percutaneous Cryoablation for the Treatment of Medically Inoperable Peripheral Lung Cancer
Brief Title: Percutaneous Cryoablation Peripheral Lung Cancer
Acronym: PCPLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Endoscope Center, Shanghai Chest Hospita, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHCHE201601
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; Percutaneous cryoablation; treatment of medically inoperable
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): Patients who are medically inoperable peripheral lung cancer will enroll in this study.They will receive percutaneous cryoablation and follow-up according to schedule.
  Interventions: Procedure: Percutaneous cryoablation

INTERVENTIONS:
Procedure: Percutaneous cryoablation — Percutaneous cryoablation

SUMMARY:
This study is focus on percutaneous cryoablation,which was for the treatment of medically inoperable Peripheral lung cancer.The patients who were agreed to attend the study will accept the operation. After the operations,they will follow up according to the plan.

DETAILED DESCRIPTION:
The patients who were agreed to attend the study conclude early stage lung cancer and solitary metastatic lung cancer.

ELIGIBILITY:
Inclusion Criteria:

medically inoperable peripheral lung cancer Diameter no more than 3cm

Exclusion Criteria:

1. Refusal of participation
2. tendency to bleed to that can't receive percutaneous cryoablation.
3. Severe cardiopulmonary dysfunction and other indications that can't receive percutaneous cryoablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years

SECONDARY OUTCOMES:
OS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sun jiayuan, MD, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Tian J, Zhao L, Wu B, Kacher DS, Ma X, Liu S, Ren C, Xiao YY. CT-guided conformal cryoablation for peripheral NSCLC: initial experience. Eur J Radiol. 2012 Nov;81(11):3354-62. doi: 10.1016/j.ejrad.2012.04.035. Epub 2012 May 23. PMID 22626572
- [Background] Kawamura M, Izumi Y, Tsukada N, Asakura K, Sugiura H, Yashiro H, Nakano K, Nakatsuka S, Kuribayashi S, Kobayashi K. Percutaneous cryoablation of small pulmonary malignant tumors under computed tomographic guidance with local anesthesia for nonsurgical candidates. J Thorac Cardiovasc Surg. 2006 May;131(5):1007-13. doi: 10.1016/j.jtcvs.2005.12.051. PMID 16678583
- [Background] Yamauchi Y, Izumi Y, Kawamura M, Nakatsuka S, Yashiro H, Tsukada N, Inoue M, Asakura K, Nomori H. Percutaneous cryoablation of pulmonary metastases from colorectal cancer. PLoS One. 2011;6(11):e27086. doi: 10.1371/journal.pone.0027086. Epub 2011 Nov 9. PMID 22096520
- [Result] Yamauchi Y, Izumi Y, Hashimoto K, Yashiro H, Inoue M, Nakatsuka S, Goto T, Anraku M, Ohtsuka T, Kohno M, Kawamura M, Nomori H. Percutaneous cryoablation for the treatment of medically inoperable stage I non-small cell lung cancer. PLoS One. 2012;7(3):e33223. doi: 10.1371/journal.pone.0033223. Epub 2012 Mar 8. PMID 22413004